CLINICAL TRIAL: NCT00182039
Title: Perioperative Ischemic Evaluation Study (POISE) Trial
Brief Title: POISE Trial: Perioperative Ischemic Evaluation Study
Acronym: POISE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Please see detailed description for reason why study was terminated.
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); National Health and Medical Research Council, Australia (Other); British Heart Foundation (Other); AstraZeneca (Industry)
Responsible Party: Dr. P.J. Devereaux, McMaster University
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MCT-50851-CT; ISRCTN17233551
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2008-04-11 (Estimated); Status verified 2008-01

CONDITIONS: Cardiovascular Diseases
Keywords: randomized controlled trial; blinded; noncardiac surgery; cardiovascular events
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): metoprolol
  Interventions: Drug: Metoprolol controlled release (CR)
- B (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metoprolol controlled release (CR) — Patients received the first dose of the study drug (i.e., oral metoprolol CR or matching placebo 100 mg) 2-4 hours prior to surgery. Administration of the study drug at each dosing time required a patient to have a heart rate ≥ 50 beats per minute (bpm) and a systolic blood pressure (SBP) ≥ 100 mmHg. If the patient's heart rate was ≥ 80 bpm and their SBP ≥ 100 mmHg at any time during the first 6 hours after surgery, the patient received their first postoperative dose (i.e., 100 mg of the study drug) orally. Patients who did not receive the study drug during the first 6 hours after surgery received 100 mg of the study drug orally at 6 hours after surgery. Twelve hours after the first postoperative dose patients started taking oral metoprolol CR or placebo 200 mg daily for 30 days.
  Arms: A
Drug: Placebo — Patients received the first dose of the study drug (i.e., oral metoprolol CR or matching placebo 100 mg) 2-4 hours prior to surgery. Administration of the study drug at each dosing time required a patient to have a heart rate ≥ 50 beats per minute (bpm) and a systolic blood pressure (SBP) ≥ 100 mmHg. If the patient's heart rate was ≥ 80 bpm and their SBP ≥ 100 mmHg at any time during the first 6 hours after surgery, the patient received their first postoperative dose (i.e., 100 mg of the study drug) orally. Patients who did not receive the study drug during the first 6 hours after surgery received 100 mg of the study drug orally at 6 hours after surgery. Twelve hours after the first postoperative dose patients started taking oral metoprolol CR or placebo 200 mg daily for 30 days.
  Arms: B

SUMMARY:
This trial will evaluate the ability of metoprolol (a beta-blocker drug) to prevent heart attacks and deaths around the time of surgery.

DETAILED DESCRIPTION:
The POISE Trial is a large multi-centre, blinded, randomized controlled group trial of metoprolol vs placebo in 10,000 at risk patients undergoing noncardiac surgery. The POISE Trial will determine the impact of perioperative administration of metoprolol on cardiovascular events (defined as cardiovascular death, nonfatal myocardial infarction, or nonfatal cardiac arrest) during the 30 day post-operative period in at risk patients undergoing noncardiac surgery.

Assuming a control group event rate of 6% for our primary outcome, we determined randomization of 8000 patients would provide 85% power and 10,000 patients 92% power to detect a relative risk reduction of 25% (two-sided alpha = 0.05). We set a goal to randomize 10,000 patients recognizing that we would have adequate power if we randomized 8000 patients. Without knowledge of the trial results and knowing that we had randomized more than 8000 patients and had a higher than predicted event rate, the Operations Committee decided to terminate recruitment on July 31, 2007 primarily because the remaining study drug expired in September 2007.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing noncardiac surgery
* ≥ 45 years of age; either sex.
* Have an expected length of stay ≥ 24 hours
* Fulfill any one of the following 6 criteria:

  * coronary artery disease;
  * peripheral vascular disease;
  * history of stroke due to atherothrombotic disease;
  * hospitalization for congestive heart failure within 3 years of randomization;
  * undergoing major vascular surgery; OR
  * any 3 of the following 7 criteria: scheduled for high risk surgery (i.e. intraperitoneal or intrathoracic); emergency/urgent surgery; any history of congestive heart failure; history of a transient ischemic attack (TIA); diabetes and currently on an oral hypoglycemic agent or insulin therapy; preoperative serum creatinine > 175 µmol/L (> 2.0 mg/dl); or age > 70 years.

Exclusion Criteria:

* Contraindication to metoprolol including any of the following: significant bradycardia (heart rate < 50 beats per minute); second or third degree heart block without a pacemaker; asthma that has been active within the last decade; and history of chronic obstructive pulmonary disease (COPD) with bronchospasm on pulmonary function tests.
* Clinical plan to use a beta-blocker preoperatively or during the first 30 postoperative days
* Prior adverse reaction to a beta-blocker
* Coronary artery bypass graft (CABG) surgery with complete revascularization in the preceding 5 years and no evidence of cardiac ischemia since the CABG surgery
* Patients undergoing low risk surgical procedures (potential examples include transurethral procedures [transurethral prostatectomies (TURPs), stone baskets, etc.], ophthalmologic procedures under topical or regional anesthesia [cornea transplants, cataract surgery, etc.], and surgeries with limited physiological stresses [digital re-implantation, nerve repairs, etc.] )
* Concurrent use of verapamil
* Prior enrollment in this trial

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8351 (Actual)
Dates: Start 2002-10; Primary Completion 2007-07 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
major cardiovascular events (defined as cardiovascular death, nonfatal myocardial infarction, or nonfatal cardiac arrest) | 30 days

SECONDARY OUTCOMES:
clinically significant atrial fibrillation rehospitalization for cardiac reasons | 30 days and 1 year
nonfatal myocardial infarction | 30 days and 1 year
nonfatal cardiac arrest | 30 days and 1 year
cardiovascular death | 30 days and 1 year
total mortality | 30 days and 1 year
revascularization procedures (i.e. coronary artery bypass surgery and percutaneous transluminal coronary angioplasty) | 30 days and 1 year
congestive heart failure | 30 days and 1 year
clinically significant bradycardia | 30 days
clinically significant hypotension | 30 days
nonfatal stroke | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: P.J. Devereaux, MD, Principal Investigator — McMaster University; Homer Yang, MD, Principal Investigator — University of Ottawa
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

REFERENCES:
- [Background] POISE Trial Investigators; Devereaux PJ, Yang H, Guyatt GH, Leslie K, Villar JC, Monteri VM, Choi P, Giles JW, Yusuf S. Rationale, design, and organization of the PeriOperative ISchemic Evaluation (POISE) trial: a randomized controlled trial of metoprolol versus placebo in patients undergoing noncardiac surgery. Am Heart J. 2006 Aug;152(2):223-30. doi: 10.1016/j.ahj.2006.05.019. PMID 16875901
- [Derived] Devereaux PJ, Xavier D, Pogue J, Guyatt G, Sigamani A, Garutti I, Leslie K, Rao-Melacini P, Chrolavicius S, Yang H, Macdonald C, Avezum A, Lanthier L, Hu W, Yusuf S; POISE (PeriOperative ISchemic Evaluation) Investigators. Characteristics and short-term prognosis of perioperative myocardial infarction in patients undergoing noncardiac surgery: a cohort study. Ann Intern Med. 2011 Apr 19;154(8):523-8. doi: 10.7326/0003-4819-154-8-201104190-00003. PMID 21502650
- [Derived] POISE Study Group; Devereaux PJ, Yang H, Yusuf S, Guyatt G, Leslie K, Villar JC, Xavier D, Chrolavicius S, Greenspan L, Pogue J, Pais P, Liu L, Xu S, Malaga G, Avezum A, Chan M, Montori VM, Jacka M, Choi P. Effects of extended-release metoprolol succinate in patients undergoing non-cardiac surgery (POISE trial): a randomised controlled trial. Lancet. 2008 May 31;371(9627):1839-47. doi: 10.1016/S0140-6736(08)60601-7. Epub 2008 May 12. PMID 18479744